CLINICAL TRIAL: NCT03470220
Title: The Role of Ultrasound in Cholecystitis
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Camilla Gustafsson, M.D. Principal Investigator, Karolinska Institutet
Other Study IDs: 2017/1222-31/2
Record Dates: First submitted 2017-11-28; First posted 2018-03-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound: All included patients will be examined with ultrasound

SUMMARY:
The aim of this study is:

1. To describe the natural course of acute cholecystitis, by performing repeated ultrasound examinations from day of admission to hospital until day of surgery or discharge.
2. To investigate if there is anything in the ultrasound picture that can predict a difficult operation.

Patients will be prospectively enrolled. The ultrasound picture (ultrasound variables: gallbladder volume, gallbladder wall thickness, and presence of oedema in the gallbladder wall), will be compared to clinical variables (tenderness in right upper quadrant, WBC, CRP and temperature) and to the time (hours) from onset of symptoms. Statistical analyses will be made to see if statistically significant, and clinically relevant, associations between variables exist.

Furthermore, for participants receiving acute surgery, an upper GI surgeon will evaluate the operation as easy, intermediate or difficult. In extension, investigators will look at associations between difficult surgery and all the variables previously mentioned (both ultrasound variables, clinical variables and time).

DETAILED DESCRIPTION:
Patients admitted to Stockholm South General Hospital's Surgery Department, with a confirmed diagnosis of acute cholecystitis (according to the Tokyo Guidelines 2013) will be considered eligible for the study and asked to participate. Informed consent will be obtained from all participants. Participants will be examined with ultrasound of the gallbladder daily, while receiving regular care for acute cholecystitis, which means either waiting for acute surgery or being treated conservatively for as long as inpatient care is needed.

The ultrasound examinations will be performed by a radiologist or a specialised certified ultrasound trained nurse as well as by an ultrasound trained surgeon. Measures of gallbladder volume (measured in cm3), gallbladder wall thickness (measured in mm:s) and presence of oedema in the gallbladder wall (noted as a binomial variable 'yes/no') are recorded in a case report form (no.1) together with body temperature, labs and information about onset of symptoms.

The operating surgeon (a specialist in surgery) will evaluate the operation and grade it from easy to difficult and fill in a case report form (no.2).

Data will be collected from the forms and analysed using a regression model (generalised estimated equation or a mixed model).

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystitis according to the Tokyo Guidelines 2013 criteria

Exclusion Criteria:

* Difficulties to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital, with confirmed acute cholecystitis according to the Tokyo Guidelines 2013 will be asked to participate in the study
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Does the gallbladder wall thickness in acute cholecystitis change over time? | Through study completion, one year
  Measurement of the gallbladder wall thickness in mm will be measured daily. Association between the gallbladder wall thickness and time from onset of symptoms (hours) will be analyzed.

SECONDARY OUTCOMES:
Does the gallbladder volume in acute cholecystitis change over time? | Through study completion, one year
  Measurement of the gallbladder volume, in cm3 will be measured daily. Association between the gallbladder volume and time from onset of symptoms (hours) will be analyzed.
Does the presence of oedema in the gallbladder wall change over time? | Through study completion, one year
  The presence of oedema in the gallbladder wall will be examined and noted daily.

OTHER OUTCOMES:
Does any of the ultrasound variables contribute to predict difficult surgery in acute cholecystitis? | Through study completion, one year
  Patients with acute cholecystitis who undergo surgery at the same admission will be included for further analysis.
  The operating surgeon (a specialist in general surgery) will classify the operation as easy, intermediate or difficult.
  Associations between difficult surgery, all the above listed variables and time from onset of symptoms will be calculated using a regression model (GEE or mixed model).

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sonden, Docent, Study Director — Karolinska Instistutet Södersjukhuset
Locations (1):
- Södersjukhuset, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Yokoe M, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Gomi H, Pitt HA, Garden OJ, Kiriyama S, Hata J, Gabata T, Yoshida M, Miura F, Okamoto K, Tsuyuguchi T, Itoi T, Yamashita Y, Dervenis C, Chan AC, Lau WY, Supe AN, Belli G, Hilvano SC, Liau KH, Kim MH, Kim SW, Ker CG; Tokyo Guidelines Revision Committee. TG13 diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):35-46. doi: 10.1007/s00534-012-0568-9. PMID 23340953
- [Background] Kiriyama S, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Yokoe M, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Gomi H, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF, Dervenis C, Chan AC, Supe AN, Liau KH, Kim MH, Kim SW; Tokyo Guidelines Revision Committee. TG13 guidelines for diagnosis and severity grading of acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):24-34. doi: 10.1007/s00534-012-0561-3. PMID 23307001
- [Background] Takada T, Strasberg SM, Solomkin JS, Pitt HA, Gomi H, Yoshida M, Mayumi T, Miura F, Gouma DJ, Garden OJ, Buchler MW, Kiriyama S, Yokoe M, Kimura Y, Tsuyuguchi T, Itoi T, Gabata T, Higuchi R, Okamoto K, Hata J, Murata A, Kusachi S, Windsor JA, Supe AN, Lee S, Chen XP, Yamashita Y, Hirata K, Inui K, Sumiyama Y; Tokyo Guidelines Revision Committee. TG13: Updated Tokyo Guidelines for the management of acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):1-7. doi: 10.1007/s00534-012-0566-y. PMID 23307006